CLINICAL TRIAL: NCT00766454
Title: Metabolic Genotypes and Oncogenic Damage in Breast Cancer
Brief Title: Studying Urine and Blood Samples in Women With Newly Diagnosed Breast Cancer
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000573065; P30CA012197 (NIH); CCCWFU-98298; CCCWFU-BG98-278
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: mutation analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: medical chart review
Other: questionnaire administration
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Studying samples of urine and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This study is looking at urine and blood samples in women with newly diagnosed breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the association between the genotype for 4 metabolic enzymes (e.g., CYP1A1, GSTM, GSTT, and GSTP) in women with newly diagnosed breast cancer that play key roles in the metabolism of environmental human carcinogens and the risk of breast cancer development.

OUTLINE: Urine and blood samples are collected for DNA, mutation, and polymorphism analysis. The biological samples may be stored and used for future research.

Patients complete a Baseline Questionnaire to collect basic risk/exposure information, including demographic factors (e.g., age, weight, height, and body mass index), menstrual/reproductive history, medical history, medication use, smoking history, alcohol consumption, exposure to chest x-ray, and family history of breast cancer in first-degree relatives. Patients also complete a Second Hand Smoke Questionnaire to collect information on cigarette smoking history and second hand smoke exposure and a Food Frequency Questionnaire to collect information on the frequency of use of specific fruits and vegetables (e.g., cruciferous vegetables) and to estimate usual dietary intake of 33 nutrients during the past year (e.g., total fat, saturated fat, oleic fat, linoleic fat, carbohydrates, protein, vitamins [e.g., A, B1, B2, niacin, B6, folate, C, and E], minerals [e.g., calcium, magnesium, iron, and zinc], electrolytes [e.g., sodium and potassium], and dietary fiber). Patients' medical charts are also reviewed to collect information on age, gender, ethnic background, medical history, and medical care.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer
* Planning to undergo a diagnostic biopsy or surgery
* Must have tumor tissue available
* Hormone receptor status not specified
* More than 6 months since prior chemotherapy or radiotherapy
* Pre- or post-menopausal

Exclusion Criteria:

-Psychiatric history that would preclude giving informed consent

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those with newly diagnosed breast cancer who are planning to undergo a diagnostic biopsy or surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1104 (Actual)
Dates: Start 1998-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Association between the genotype for 4 metabolic enzymes (e.g., CYP1A1, GSTM, GSTT, and GSTP) that play key roles in the metabolism of environmental human carcinogens and the risk of breast cancer development | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Akman, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States